CLINICAL TRIAL: NCT05400811
Title: Prospective, Randomised, DBPC, Double-dummy, Multicenter CT of Efficacy and Safety With IT in Patients With Controlled Mild to Moderate Allergic Asthma and Rhinitis/Rhinoconjunctivitis, Allergic to D. Pteronyssinus and/or D. Farinae.
Brief Title: Efficacy and Safety Evaluation for the Treatment of HDM Induced Allergic Asthma and Rhinitis/Rhinoconjunctivitis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Inmunotek S.L. (Industry)
Collaborators: BioClever 2005 S.L. (Other); NTS hub S.L (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MM09-SIT-040
Record Dates: First submitted 2022-05-27; First posted 2022-06-02 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-04

CONDITIONS: House Dust Mite Allergy; Perennial Allergic Rhinitis; Allergic Rhinoconjunctivitis; Allergic Asthma
Keywords: Rhinitis/ Rhinoconjunctivitis; Allergy; Immunotherapy; Mild to moderate asthma
MeSH Terms: conditions — Dust Mite Allergy; Rhinitis, Allergic, Perennial; Hypersensitivity

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, placebo-controlled, double-blind, double-dummy, multi-center trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: During the trial, both the investigator and the included subjects will be unaware of the treatment each subject is receiving.
  The person in charge of data analysis will also not know the treatment assigned to each subject until the database has been closed.
  Neither the subject nor the investigator knows what treatment each subject is receiving, all the trial medication is identical in terms of outer packaging and appearance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group I: MM09 allergoid-mannan conjugates SC (3.000 UTm/mL) + sublingual placebo (Experimental): Mixture of allergen extracts of Dermatophagoides pteronyssinus and Dermatophagoides farinae conjugated to mannan at 3,000 UTm/mL subcutaneous immunotherapy + sublingual placebo.
  Subcutaneous active treatment will be administered once a month for 12 months. Sublingual placebo will be administered daily (2 subsequent administrations) for 12 months.
  Interventions: Biological: MM09 allergoid-mannan conjugates subcutaneous (3.000 UTm/mL); Biological: Placebo sublingual
- Group II: MM09 allergoid-mannan conjugates SL (3.000 UTm/mL) + subcutaneous placebo (Experimental): Mixture of allergen extracts of Dermatophagoides pteronyssinus and Dermatophagoides farinae conjugated to mannan sublingual immunotherapy at 3.000 UTm/mL + subcutaneous placebo.
  Sublingual active treatment will be administered daily (2 subsequent administrations) for 12 months.
  Subcutaneous placebo will be administered once a month for 12 months.
  Interventions: Biological: MM09 allergoid-mannan conjugates Sublingual (3.000 UTm/mL); Biological: Placebo subcutaneous
- Group III: MM09 allergoid-mannan conjugates SL (9.000 UTm/mL) + subcutaneous placebo (Experimental): Mixture of allergen extracts of Dermatophagoides pteronyssinus and Dermatophagoides farinae conjugated to mannan sublingual immunotherapy at 9.000 UTm/mL + subcutaneous placebo.
  Sublingual active treatment will be administered daily (2 subsequent administrations) for 12 months.
  Subcutaneous placebo will be administered once a month for 12 months.
  Interventions: Biological: MM09 allergoid-mannan conjugates Sublingual (9.000 UTm/mL); Biological: Placebo subcutaneous
- Group IV: Placebo (Placebo Comparator): Mixture of sublingual placebo + subcutaneous placebo. Sublingual placebo will be administered daily (2 subsequent administrations) for 12 months.
  Subcutaneous placebo will be administered once a month for 12 months
  Interventions: Biological: Placebo subcutaneous; Biological: Placebo sublingual

INTERVENTIONS:
Biological: MM09 allergoid-mannan conjugates subcutaneous (3.000 UTm/mL) — Mixture of allergen extracts of Dermatophagoides pteronyssinus and Dermatophagoides farinae conjugated to mannan at 3.000 UTm/mL for subcutaneous administration.
  Arms: Group I: MM09 allergoid-mannan conjugates SC (3.000 UTm/mL) + sublingual placebo
Biological: MM09 allergoid-mannan conjugates Sublingual (3.000 UTm/mL) — Mixture of allergen extracts of Dermatophagoides pteronyssinus and Dermatophagoides farinae conjugated to mannan at 3.000 UTm/mL for sublingual administration.
  Arms: Group II: MM09 allergoid-mannan conjugates SL (3.000 UTm/mL) + subcutaneous placebo
Biological: MM09 allergoid-mannan conjugates Sublingual (9.000 UTm/mL) — Mixture of allergen extracts of Dermatophagoides pteronyssinus and Dermatophagoides farinae conjugated to mannan at 9.000 UTm/mL for sublingual administration.
  Arms: Group III: MM09 allergoid-mannan conjugates SL (9.000 UTm/mL) + subcutaneous placebo
Biological: Placebo subcutaneous — The same solution, presentation, method of administration, frequency, and duration as the active treatment, but without active ingredients.
  Arms: Group II: MM09 allergoid-mannan conjugates SL (3.000 UTm/mL) + subcutaneous placebo; Group III: MM09 allergoid-mannan conjugates SL (9.000 UTm/mL) + subcutaneous placebo; Group IV: Placebo
Biological: Placebo sublingual — The same solution, presentation, method of administration, frequency, and duration as the active treatment, but without active ingredients.
  Arms: Group I: MM09 allergoid-mannan conjugates SC (3.000 UTm/mL) + sublingual placebo; Group IV: Placebo

SUMMARY:
Prospective, randomized, placebo-controlled, multicenter of 3 active treatment groups, compared to 1 placebo group, for the determination of the efficacy and safety of subcutaneous immunotherapy in patients with mild to moderate asthma and rhinitis/rhinoconjunctivitis (intermittent or persistent) allergic to Dermatophagoides pteronyssinus and/or Dermatophagoides farinae.

DETAILED DESCRIPTION:
Prospective multicenter randomized double-dummy clinical trial of three active treatment groups compared to one placebo group. The principal objective of the clinical trial is the determination of the efficacy and safety of subcutaneous immunotherapy in patients with mild to moderate asthma and rhinitis/rhinoconjunctivitis (intermittent or persistent) allergic to Dermatophagoides pteronyssinus and/or Dermatophagoides farinae.

The primary efficacy endpoint will be the symptom score and medication consumption required for the control of asthma and rhinitis/rhinoconjunctivitis symptoms.

The study design consists of 3 active treatment groups and one placebo group. The trial population will include 400 subjects between the age of 12 and 60 years that will receive the treatment during 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated Informed Consent Form (ICF).
2. Female or male aged 12 to 60 years, both included.
3. Confirmed clinical history of inhalation allergy (mild-moderate controlled intermittent or persistent asthma according to the definition of GEMA 5.0 and GINA 2020 and intermittent or persistent rhinitis / rhinoconjunctivitis according to the ARIA classification, caused by Dermatophagoides pteronyssinus and / or Dermatophagoides farinae). The asthma diagnosis will be valid up to 24 months prior to signing the informed consent.
4. Positive skin prick test (wheal major diameter ≥ 5 mm) to a standardized allergen extract of Dermatophagoides pteronyssinus and/or Dermatophagoides farinae.
5. Specific IgE against a complete extract of D. pteronyssinus and/or D. farinae or any of the molecular components of allergenic sources with a value ≥ 3.5 kU/L.
6. Women of childbearing age must have a urine pregnancy test negative result before enrolling the study.
7. Women of childbearing age must commit to using an adequate contraception method.
8. Capable of complying with dosage regimen.
9. Owning a smartphone to register symptoms and medication consumption.
10. A negative skin prick test to other aeroallergens with specific IgE < 3.5 kU/L with no clinical relevance.

Exclusion Criteria:

1. Previous immunotherapy to any of the tested allergen during the last 5 years or any desensitization process in the last 2 years (ITO, milk, egg, ...) or currently receiving immunotherapy with any other allergen.
2. Positive skin prick test to other aeroallergens, except for intermittent symptoms due to temporary exposition to dander.
3. Those cases in which AIT would be a contraindication according to the criteria of European Allergy and Clinical Immunology Immunotherapy Subcommittee.
4. Uncontrolled or severe asthma and/or FEV1 <70% despite pharmacological treatment by the time of enrolment.
5. Intake of β-blockers.
6. Use of immunosuppressive or biological drug.
7. Unstable patients by the time of enrolment (acute exacerbation asthma, respiratory infection, fever, acute pruritus, etc).
8. Patients who have suffered chronic urticaria during the last 2 years, severe anaphylaxis, or family history of angioedema.
9. Having any contraindication for the use of adrenaline (hyperthyroidism, heart disease, high blood pressure).
10. Other severe diseases not related to allergic asthma or rhinitis that could interfere in the study treatment or the follow-up (epilepsy, psychomotor agitation, diabetes, malformations, nephropathy) according to medical criteria.
11. Autoimmune diseases (thyroiditis, lupus, etc.), tumoral diseases or immunodeficiencies.
12. Participants that the investigator believes could not comply with the study protocol or have serious psychiatric disorders.
13. Known allergy to any of the ingredients of the study medication except for mites.
14. Lower respiratory tract diseases different from asthma as bronchiectasis or chronic obstructive pulmonary disease.
15. Breast-feeding or pregnant women.
16. Being immediate family of the investigator.
17. Concurrent participation in other clinical trials or prior participation within 30 days prior to inclusion.
18. History of serious systemic reactions, including food, Hymenoptera venom, medications, etc.

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
CSMS: Combined Symptoms and Medication Score | 12 months
  Evaluation of the number of symptoms and the consumption of medication necessary for the control of such symptoms in asthma and rhinitis / rhinoconjunctivitis of each subject during the trial, of the groups with each other and with respect to placebo.
  - The endpoint for each asthma and rhinitis / rhinoconjunctivitis symptom will be as follows: 0 = No symptoms; 1 = Mild; 2 = Moderate; 3 = Severe
  Total daily symptom score = 0-3
  The asthma medication will be scored based on the therapeutic step in which drugs are included in the GEMA 5 guide.
  The rhinitis / rhinoconjunctivitis medication score: 0 = No medication; 1 = oral or topical (eyes or nose) non-sedative H1 antihistamines (H1A); 2 = intranasal corticosteroids (INS) with / without H1A; 3 = oral corticosteroids with/without (INS), with/without H1A Total daily medication score = 0-3

SECONDARY OUTCOMES:
Asthma symptom-free days | 12 months
  Number of days that subjects have no symptoms related to asthma
Rhinitis / rhinoconjunctivitis symptom-free days | 12 months
  Number of days that subjects have no symptom related to rhinitis / rhinoconjunctivitis.
Asthma medication-free days | 12 months
  Number of days that subjects need no medication for treatment of asthma.
Rhinitis / rhinoconjunctivitis medication-free days | 12 months
  Number of days that subjects need no medication for treatment of Rhinitis / rhinoconjunctivitis.
Respiratory function_FEV1 | Baseline, month 6, month 12
  Measurement of Forced Expiratory Volume in 1 Second (FEV1) %
Respiratory function_PEF | Baseline, month 6, month 12
  Peak Expiratory Flow (PEF) [velocity]
Asthmatic exacerbations | 12 months
  Time elapsed until the first appearance of asthmatic exacerbations, number, duration and severity.
Clinical benefit | 12 months
  Time to onset of clinical benefit
Immunological parameters | 12 months
  Analyses of total and specific IgE, specific IgE index / total IgE, specific IgG4 and Anti-Saccharomyces cerevisiae (ASCA) IgA&IgG.
Quality of life associated with asthma (AQLQ) | 12 months
  The quality of life associated with asthma will be measured using the Asthma Quality of Life Questionnaire (AQLQ).
  AQLQ consists of 32 items and 4 domains (limitations in activities, symptoms, emotional and environmental). Each item is scored from 1=no impairment to 7=severe impairment.
Quality of life associated with rhinoconjunctivitis (RQLQ) | Baseline, month 6, month 12
  The quality of life associated with rhinoconjunctivitis will be measured using the Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ).
  RQLQ it consists of 28 items (questions) and 7 domains (Activities, sleep, general symptoms, practical problems, nose symptoms, eye and emotional symptoms).
  The score of each item for all domains, except for the emotional one, ranges from "0=Nothing bothered me" to "6=It has bothered me a lot". The emotional domain score ranges from "0=Never" to "6=Always".
Questionnaire for asthma control (ACQ) | 12 months
  Asthma control will be measured following the ACQ questionnaire.
  The ACQ questionnaire consists of 7 questions (ACQ-7) or 6 questions (ACQ-6). In questions 1-6, patients recall their experience during the last 7 days and answer using a scale of 7 points (from "0 = fully controlled" to "6 = extremely poorly controlled"). The seventh question, which refers to the% FEV1 of the reference value, must be completed by an employee of the site. The questionnaire score is the mean of the 7 responses (ACQ-7) or 6 responses (ACQ-6).
  The interpretation of the scores is as follows:
  Less than or equal to 0.75: Adequate control of asthma From 0.75 to 1.50: Partially controlled asthma More than 1.50: Inadequate asthma control
Visual Analogue Scale (VAS) | 12 months
  Visual Analogue Scale in which the subject has to indicate in a straight line of 10 cm how he/she feels regarding to his allergy symptoms. Being left side "0 = very bad" and right side "10 = very well".
  VAS scale will also be completed by the investigator answering how he/she thinks that the patient feels.
Consumption of health resources | 12 months
  For each patient, the number of times that due to allergy symptoms has done the following will be counted:
  * have visited the family doctor
  * have made an unscheduled visit to the specialist
  * has gone to the emergency room
  * has been hospitalized
  * have needed to contact the doctor by phone
Safety parameters | 12 months
  Global rate and severity of AE per administration and per subject
Number of Local Adverse Reactions | 12 months
  Local adverse reactions are those that appear at the site of the administration. They are classified into: Immediate (it appears during the first 30 minutes from the administration of investigational product) and Late (it appears after the first 30 minutes from the administration of investigational product)
Number of Systemic Adverse Reactions | 12 months
  Systemic adverse reactions are those that appear in other parts of the body other than the site of administration.Their severity will be classified following the indications proposed by the World Allergy Organization (WAO) in 2010.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Isabel Tabar Purroy, MD. PhD, Principal Investigator — Hospital of Navarra
Locations (16):
- Spain (16):
  - Hospital Universitario de Elche, Elche, Alicante
  - Policlínica Nuestra Sra del Rosario, Ibiza Town, Balearic Islands
  - Hospital Sant Joan de Déu, Esplugues de Llobregat, Barcelona
  - Hospital de Terrassa, Terrassa, Barcelona
  - Hospital Universitario de Navarra, Pamplona, Navarre
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Hospital Universitario A Coruña, A Coruña
  - Hospital General Universitario de Alicante, Alicante
  - Centro Médico Quiron Salud Alicante, Alicante
  - Hopital Quirón Salud Málaga, Málaga
  - Clinica del Dr.Pérez Estrada Cornejo, Málaga
  - Hospital Universitario Regional de Málaga, Málaga
  - Clínica RUSADIR, Melilla
  - Complexo Hospitalario Universitario de Pontevedra, Pontevedra
  - Hospital Univeristario y Politécnico La Fe, Valencia
  - Hospital Universitario de la Plana, Vila-real

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benito-Villalvilla C, Soria I, Subiza JL, Palomares O. Novel vaccines targeting dendritic cells by coupling allergoids to mannan. Allergo J Int. 2018;27(8):256-262. doi: 10.1007/s40629-018-0069-8. Epub 2018 May 18. PMID 30546997
- [Background] Sirvent S, Soria I, Cirauqui C, Cases B, Manzano AI, Diez-Rivero CM, Reche PA, Lopez-Relano J, Martinez-Naves E, Canada FJ, Jimenez-Barbero J, Subiza J, Casanovas M, Fernandez-Caldas E, Subiza JL, Palomares O. Novel vaccines targeting dendritic cells by coupling allergoids to nonoxidized mannan enhance allergen uptake and induce functional regulatory T cells through programmed death ligand 1. J Allergy Clin Immunol. 2016 Aug;138(2):558-567.e11. doi: 10.1016/j.jaci.2016.02.029. Epub 2016 Apr 13. PMID 27177779
- [Background] Manzano AI, Javier Canada F, Cases B, Sirvent S, Soria I, Palomares O, Fernandez-Caldas E, Casanovas M, Jimenez-Barbero J, Subiza JL. Structural studies of novel glycoconjugates from polymerized allergens (allergoids) and mannans as allergy vaccines. Glycoconj J. 2016 Feb;33(1):93-101. doi: 10.1007/s10719-015-9640-4. Epub 2015 Nov 25. PMID 26603537
- [Background] Soria I, Lopez-Relano J, Vinuela M, Tudela JI, Angelina A, Benito-Villalvilla C, Diez-Rivero CM, Cases B, Manzano AI, Fernandez-Caldas E, Casanovas M, Palomares O, Subiza JL. Oral myeloid cells uptake allergoids coupled to mannan driving Th1/Treg responses upon sublingual delivery in mice. Allergy. 2018 Apr;73(4):875-884. doi: 10.1111/all.13396. Epub 2018 Jan 31. PMID 29319882
- [Background] Soria I, Alvarez J, Manzano AI, Lopez-Relano J, Cases B, Mas-Fontao A, Canada FJ, Fernandez-Caldas E, Casanovas M, Jimenez-Barbero J, Palomares O, Vinals-Florez LM, Subiza JL. Mite allergoids coupled to nonoxidized mannan from Saccharomyces cerevisae efficiently target canine dendritic cells for novel allergy immunotherapy in veterinary medicine. Vet Immunol Immunopathol. 2017 Aug;190:65-72. doi: 10.1016/j.vetimm.2017.07.004. Epub 2017 Jul 23. PMID 28778325
- [Background] Gonzalez JL, Zalve V, Fernandez-Caldas E, Cases B, Subiza JL, Casanovas M. A pilot study of immunotherapy in dogs with atopic dermatitis using a mannan-Dermatophagoides farinae allergoid targeting dendritic cells. Vet Dermatol. 2018 Oct;29(5):449-e152. doi: 10.1111/vde.12679. PMID 30183126